CLINICAL TRIAL: NCT06047691
Title: Randomized Controlled Trial of Intensive Multi-Couple Therapy for PTSD Versus Relationship Education in Military Couples
Brief Title: Intensive Multi-Couple Therapy for PTSD Versus Relationship Education in Military Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); University of Denver (Other); Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Steffany J Fredman, Ph.D., Associate Professor of Human Development and Family Studies and Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SITE00001245
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with parallel group design
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be blinded as to participant treatment condition during follow-up assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abbreviated, Intensive, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy for PTSD (Experimental): AIM-CBCT for PTSD is an abbreviated, intensive, multi-couple group version of cognitive-behavioral conjoint therapy for PTSD, an evidence-based treatment for PTSD delivered in a conjoint format.
  Interventions: Behavioral: Abbreviated, Intensive, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy for PTSD
- Prevention and Relationship Education Program (Active Comparator): PREP is an evidence-based relationship education program delivered in a multi-couple group format.
  Interventions: Behavioral: Prevention and Relationship Education Program

INTERVENTIONS:
Behavioral: Abbreviated, Intensive, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy for PTSD — Approximately 12 hours of programming delivered over 2 consecutive days in a multi-couple group retreat format. Couples are provided with psychoeducation about PTSD and relationship functioning and are taught cognitive and behavioral skills to address the manifestation of PTSD in the couple relationship. Couples will also meet once individually with one of the group leaders 1-2 weeks before the retreat and once 1-2 weeks after the retreat.
  Arms: Abbreviated, Intensive, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy for PTSD
Behavioral: Prevention and Relationship Education Program — Approximately 12 hours of programming delivered over 2 consecutive days in a multi-couple group retreat format.The content of PREP and workshop experiences focuses on helping couples communicate effectively, manage conflict without harming their relationship, preserve and act on commitment, improve relationship decision-making, increase understanding of differences between partners, and protect positive connections between partners. Approximately 12 hours of PREP content will be delivered over 2 consecutive days in a multi-couple group retreat format. Couples will also meet once individually with one of the group leaders 1-2 weeks before the retreat and will check in with a member of the study staff 1-2 weeks after the retreat.
  Arms: Prevention and Relationship Education Program

SUMMARY:
The goal of this clinical trial is to test an abbreviated, intensive, multi-couple group version of cognitive-behavioral conjoint therapy for PTSD (AIM-CBCT for PTSD) in an active military and veteran population. The main questions it aims to answer are:

* Does AIM-CBCT for PTSD improve PTSD symptoms?
* Does AIM-CBCT for PTSD improve associated symptoms (e.g., depression), romantic partner distress, and couple relationship satisfaction?

Participants will participate in a two-day retreat in which they are taught and practice skills to decrease PTSD symptoms and enhance their relationships. Researchers will compare AIM-CBCT for PTSD to the Prevention and Relationship Education Program (PREP) to determine whether it is superior to an evidence-based relationship education curriculum that is also delivered in a two-day multi-couple group format.

ELIGIBILITY:
Inclusion Criteria:

* Service member or veteran and a romantic partner willing to participate.
* Couple is married or cohabiting for at least 3 months. Couple can be either different or same sex.
* Service member/veteran diagnosis of PTSD as determined by the CAPS-5.
* Each partner is at least 18 years old.
* Both partners able to speak and read English.

Exclusion Criteria:

* Either partner reports current suicidal ideation severe enough to warrant immediate attention
* Current homicide risk meriting crisis intervention for either partner
* Current and severe alcohol misuse in either partner in the past 12 weeks and/or warranting immediate intervention
* Recent (past month) manic episode or psychotic disorder symptoms in either partner
* Evidence of a moderate or severe traumatic brain injury or other cognitive impairment in either partner
* Couple is separated or have taken steps to dissolve their relationship
* Either partner is currently participating in evidence-based treatment for PTSD (e.g., Prolonged Exposure, Cognitive Processing Therapy, Present-Centered Therapy for PTSD, Eye Movement Desensitization and Reprocessing, Cognitive-Behavioral Conjoint Therapy for PTSD, or Structured Approach Therapy).
* Evidence or admission of severe intimate aggression as indicated by a "yes" endorsement to the one-question Screen for Conflict Question by either partner occurring within the past 6-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Interviewer ratings of posttraumatic stress disorder (PTSD) symptoms identified in the Diagnostic and Statistical Manual for Mental Disorders, Fifth Edition. Scores range from 0-80, with higher scores indicating more severe PTSD symptoms.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Participant's self-report of posttraumatic stress disorder (PTSD) symptoms identified in the Diagnostic and Statistical Manual for Mental Disorders, Fifth Edition. Scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Patient Health Questionnaire-9 | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Self-reported depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depressive symptom severity.
Generalized Anxiety Disorder-Screener | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Self-reported general anxiety symptoms. Scores range from 0 to 21, with higher scores indicating greater anxiety.
Dimensions of Anger Reactions-5 | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Self-reported anger symptoms. Scores range from 5 to 25, with higher scores indicating greater anger.
Couples Satisfaction Index-32 | baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Self-reported relationship satisfaction. Scores range from 0 to 161, with higher scores indicating higher relationship satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Steffany J Fredman, Ph.D., Principal Investigator — Penn State University
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No